CLINICAL TRIAL: NCT03823131
Title: The Trifecta Study: Optimizing Antitumor Immunity Using Plasmid Electroporation, Pembrolizumab, and Epacadostat
Brief Title: Optimizing Antitumor Immunity Using Plasmid Electroporation, Pembrolizumab, and Epacadostat
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment Ineffective
Sponsor: Chase Heaton, MD (Other)
Collaborators: Incyte Corporation (Industry); OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Chase Heaton, MD, Asst Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 172021; NCI-2018-02901 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Unresectable Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Electroporation; Electroporation Therapies; epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Arm A: Tavo-EP, pembrolizumab, epacadostat (Experimental): Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks to up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30 minute IV infusion at a dose of 200 mg every 3 weeks. Epacadostat will be administered at the dose level determined in the dose escalation safety lead-in.
  Interventions: Device: ImmunoPulse; Drug: Epacadostat; Drug: Pembrolizumab; Drug: Tavokinogene telseplasmid
- Arm B: Tavo-EP, pembrolizumab (Experimental): Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks to up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30 minute IV infusion at a dose of 200 mg every 3 weeks.
  Interventions: Device: ImmunoPulse; Drug: Pembrolizumab; Drug: Tavokinogene telseplasmid
- Arm C: Tavo-EP, pembrolizumab, CORVax (Experimental): Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks to up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30-minute IV infusion at a dose of 200 mg every 3 weeks. CORVax will be administered at a total dose of 0.2 mg of (S) protein plasmid in 120 microliter (uL) per lesion intratumorally into a maximum of 4 lesions of at least 0.3 mm in diameter for a total plasmid dose of 0.8 mg on treatment days 1 and 29 of cycle 1 followed by electroporation of the plasmid solution in infiltrated regions. On days when both tavo and CORVax is administered to the same lesions, tavo and CORVax will each be injected into the lesion followed by electroporation.
  Interventions: Device: ImmunoPulse; Drug: Pembrolizumab; Biological: CORVax; Drug: Tavokinogene telseplasmid

INTERVENTIONS:
Device: ImmunoPulse — Intratumoral
  Other Names: Electroporation; electroporation therapy (EPT)
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
  Arms: Arm A: Tavo-EP, pembrolizumab, epacadostat
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: CORVax — Intratumoral
  Other Names: DNA-encodable coronaviral vaccine
  Arms: Arm C: Tavo-EP, pembrolizumab, CORVax
Drug: Tavokinogene telseplasmid — Intratumoral
  Other Names: Tavo-EP; DNA plasmid; plasmid IL-12 pUMVC3-hIL-12-NGVL3

SUMMARY:
This phase II trial studies how well tavokinogene telseplasmid with electroporation (tavo-EP), pembrolizumab, and epacadostat work in treating patients with squamous cell carcinoma of the head and neck that cannot be removed by surgery. Tavokinogene telseplasmid with electroporation is a gene therapy that may delay of tumor growth and which may have less toxicity than other methods of gene delivery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving tavokinogene telseplasmid with electroporation, pembrolizumab, and epacadostat may work better in treating squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Dose Escalation Safety Lead-Ins: Assess the safety of tavo-EP and pembrolizumab in combination with epacadostat (CTCAE version 4).

II. Dose Expansion: Determine whether the combination therapy in each arm increases the best overall response rate (BORR) compared with historical data for pembrolizumab monotherapy

SECONDARY OBJECTIVES:

I. Dose Expansion: Determine the durability of clinical benefits in participants treated with combination therapy in each arm, as assessed by time to progression, median progression-free survival (PFS), median overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Determine the effects of combination therapy on treated and untreated lesions by examining paired biopsy specimens for changes in inflammatory gene expression, relative proportion of effector versus regulatory T cells, evaluation of inflammatory cytokines, T-cell activation, clonality, and other hallmarks of immune activation.

II. Explore systemic markers of immune activation by examining circulating T-cell populations for changes in the frequency and effector function of short-lived effector cells and memory T cells.

III. Explore changes in functional immune responses using Elispot and other assays.

IV. To explore biomarkers that inform scientific understanding of this therapeutic treatment through analysis of specimens retained for Future Biomedical Research.

OUTLINE:

This is a multi-center, open label, 2-stage, double-arm, clinical trial in which participants in Stage 1 will receive either tavo-EP with pembrolizumab, and epacadostat (Arm A), tavo-EP and pembrolizumab (Arm B), or CORVax, tavo-EP and pembrolizumab (Arm C). Arms B and C will only open to enrollment if the treatment is determined to be effective in Arm A.

Participants will be followed at 3-month intervals for toxicity and radiographic imaging (1) until start of a new anti-cancer treatment, (2) until 30 days after documented disease progression, (3) until death, or (4) until 36 months from the initiation of treatment on study, whichever comes first. Each subject will be followed for overall survival until death, withdrawal of consent, or at the time of study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Life expectancy of at least 4 months.
* Patients must have histological or cytological diagnosis of cancer originating in the head and neck that is not amenable to surgical resection or locoregional radiation therapy with curative intent.
* At least one accessible lesion (AL) for intratumoral injection. An AL is defined as meeting the following criteria; (1) at least 0.3 cm x 0.3 cm in longest perpendicular diameters (2) in a suitable location for application of electroporation. Tumors invading the carotid artery or at other sites that the investigator believes to be at high risk of life-threatening hemorrhage should not be injected and these lesions may not be used to meet the inclusion criterion for injectable lesions.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1; at least one lesion where the longest perpendicular diameter is at least 1.0 cm by clinical measurement; or at least 1.0 cm by radiographic imaging for non-nodal lesions; at least 1.5 cm in short axis by radiographic imaging for malignant lymph nodes; If the biopsied lesions were previously irradiated, they must demonstrate either radiographic or pathological evidence of recurrent or residual disease. It is not necessary that this lesion is also an AL.
* If patient has known brain metastases, they must have stable neurologic status following local therapy (surgery or radiation) for at least 4 weeks without the use of steroids or on stable or decreasing dose of <=10 mg daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs) (patients with a history of carcinomatous meningitis are not eligible).
* Patients may have had prior chemotherapy or immunotherapy or radiation therapy. Any drug related adverse events identified during prior therapy must be well controlled (typically resolution to =< grade 1, OR resolved upon investigator review prior to initiation of this therapy.
* No systemic antineoplastic therapy may be received by the patient between the time of the biopsy and the first administration of study treatment.
* Patient must agree to any protocol mandated biopsies of tumor (deemed accessible and safe for biopsy by the investigator's assessment) and they must allow acquired tissue to be used for biomarker analysis.
* For women of childbearing potential, negative serum or urine pregnancy test within 14 days of first dose of study drug(s) and use of birth control from 30 days prior to the first study drug administration and 120 days following last administration of study drug, or for participants in Arm C, 180 days after last dose of CORVax, whichever is longer.
* Male patients must be surgically sterile or must agree to use contraception during the study and at least 120 days following the last administration of study drug, or for participants in Arm C, 180 days after last dose of CORVax, whichever is longer.

Exclusion Criteria:

* Active autoimmune disease that has required systemic treatment in past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Congestive heart failure (New York Heart Association class III to IV)
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful. Screening corrected QT (QTc) interval > 480 milliseconds is excluded. In the event that a single QTc is > 480 milliseconds, the subject may enroll if the average QTc for the 3 ECGs is < 480 milliseconds. For subjects with an intraventricular conduction delay (QRS interval > 120 milliseconds), the corrected JT (JTc) interval may be used in place of the QTc with sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. Subjects with left bundle branch block are excluded.
* Uncontrolled or clinically significant conduction abnormalities (e.g., ventricular tachycardia on anti-arrhythmics are excluded), 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block (LAFB)/right bundle branch block (RBBB) are eligible.
* Uncontrolled, symptomatic ischemia within 6 months of first dose of study treatment or known myocardial infarction in the previous six months.
* Patients with electronic pacemakers or defibrillators.
* Has history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Any other current or previous malignancy within the past 2 years that, in the opinion of the principal investigator will interfere with study-specific endpoints.
* Evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) requiring systemic therapy at time of study enrollment.
* Hepatitis B: Most nasopharyngeal cancer (NPC) patients have been infected with hepatitis B (Cancer Epidemol Biomarkers Prev. 2015. 24:1766-73, N = 711) and, therefore, the inclusion of healthy patients with a history of hepatitis B is a central part of this study. In addition, programmed cell death protein 1 (PD-1) antibodies have been proven to be safe in patients with active hepatitis and hepatocellular carcinoma (e.g. KEYNOTE 224). However, patients with hepatitis B virus (HBV) surface antigen positive (HBSAg) must have aspartate aminotransferase (AST) and total bilirubin < 1.5 x upper limit of normal (ULN) AND
* Negative HBV ribonucleic acid (RNA) polymerase chain reaction (PCR) OR
* On antivirals for HBV AND at least 8 weeks of prior anti-PD-1 antibody therapy AND no history of AST or total bilirubin levels > 1.5 x ULN due to PD-1 antibody therapy
* Hepatitis C (hepatitis C virus (HCV) RNA (qualitative) is detected).
* Presence of a gastrointestinal condition that may affect drug absorption. Administration of epacadostat through a feeding tube is permitted.
* Patients receiving systemic steroid therapy for a chronic inflammatory condition. Topical steroids, nasal and inhaled steroids are permitted. Prednisone or equivalent =< 10 mg/day is permitted as hormone replacement; higher dosage prednisone should be stopped at least 14 days prior to course 1 day 1 (C1D1).
* Receipt of a live vaccine or live attenuated vaccine within 30 days before the first dose of study treatment. Administration of killed vaccines is allowed.
* Subjects receiving monoamine oxidase inhibitors (MAOIs) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) within the 21 days before screening.
* Any history of serotonin syndrome (SS) after receiving serotonergic drugs.
* Use of any uridine 5'-diphospho-glucuronosyltransferase 1-9 (UGT1A9) inhibitor from screening through follow-up period, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
* Known allergy or reaction to any component of study drug formulation.
* Absolute neutrophil count (ANC) < 1.0 x 10^9/L.
* Platelets < 75 x 10^9/L.
* Hemoglobin < 9 g/dL or < 5.6 mmol/L (transfusion is acceptable to meet this criterion).
* Serum creatinine >= 1.5 x institutional upper limit of normal (ULN) OR measured or calculated creatinine clearance [glomerular filtration rate can also be used in place of creatinine or creatinine clearance (CrCl)] < 50 mL/min for subjects with creatinine levels > 1.5 x institutional ULN.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x institutional ULN.
* Alkaline phosphatase > 2.5 x ULN. Note: Subjects with 1) bone metastases and gamma-glutamyl transpeptidase (GGT) < 2.5 x ULN may enroll if the alkaline phosphatase is < 5 x ULN.
* Total bilirubin above 1.5 x the institutional ULN AND conjugated bilirubin >= 2.0 x ULN.
* International normalized ratio (INR) or prothrombin time (PT) > 1.5 x ULN.
* Activated partial thromboplastin time (aPTT) > 1.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chase Heaton, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment in Arm A was terminated earlier than expected. Arms B and Arm C were never opened for enrollment.
Groups:
- Arm A: Tavo-EP, Pembrolizumab, Epacadostat: Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks, for up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30 minute IV infusion at a dose of 200 mg every 3 weeks. Epacadostat will be administered at the dose level determined in the dose escalation safety lead-in.
- Arm B: Tavo-EP, Pembrolizumab: Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks, for up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30 minute IV infusion at a dose of 200 mg every 3 weeks.
- Arm C: Tavo-EP, Pembrolizumab, CORVax: Tavo-EP will be injected intratumorally on Days 1, 5 and 8 every 6 weeks, for up to 7 accessible lesions without exceeding 20 mL per day. Injected lesions will then be electroporated using the ImmunoPulse electroporation device. Pembrolizumab will be administered by a 30-minute IV infusion at a dose of 200 mg every 3 weeks. CORVax will be administered at a total dose of 0.2 mg of (S) protein plasmid in 120 microliter (uL) per lesion intratumorally into a maximum of 4 lesions of at least 0.3 mm in diameter for a total plasmid dose of 0.8 mg on treatment days 1 and 29 of cycle 1 followed by electroporation of the plasmid solution in infiltrated regions. On days when both tavo and CORVax is administered to the same lesions, tavo and CORVax will each be injected into the lesion followed by electroporation.
Period: Overall Study
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat | Arm B: Tavo-EP, Pembrolizumab | Arm C: Tavo-EP, Pembrolizumab, CORVax
Started | 14 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety and efficacy analysis population is defined as all enrolled subjects who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat | Arm B: Tavo-EP, Pembrolizumab | Arm C: Tavo-EP, Pembrolizumab, CORVax | Total
Number analyzed (Participants) | 14 | 0 | 0 | 14
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 0 | 0 | 1
  40-49 years old | 3 | 0 | 0 | 3
  50-59 years old | 3 | 0 | 0 | 3
  60-69 years old | 4 | 0 | 0 | 4
  70-79 years old | 3 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 12 | 0 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 12 | 0 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 0 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 0 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: The best overall response (BORR) is defined as the best response recorded from the start of treatment until disease progression/recurrence. Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, Complete Response (CR) is defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is defined as having at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The combined percentage of participants relative to the total size of the All Treated Subjects population having a demonstrated best response of CR or PR, with a confirmatory scan will be reported.
Time Frame: Up to 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
percentage of participants | 0

2. Secondary Outcome: Median Months of Progression-Free Survival (PFS)
Description: Progression-free survival will be calculated as number of months from the first dosing date until the date of disease progression (i.e the date of the tumor imaging following baseline per central imaging assessment by a radiologist) or death from any cause. Per RECIST version 1.1, Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Participants who do not have documented disease progression will have their months of PFS censored on the last date of tumor assessment, or death, whichever comes first. Censoring data on date of last tumor imaging to calculate the median PFS will not occur until the overall survival data collection for all participants has been completed.
Time Frame: Up to 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
months | 1.76 [0.89 to 5.26]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival (OS) is defined as the number of months from the date of enrollment until the date of death regardless of cause, last date of follow-up, or date of study closure (if still alive), whichever comes first. Median months of overall participant survival will be reported using descriptive statistics.
Time Frame: Up to 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
months | 11.6 [1.02 to 36]

4. Secondary Outcome: Median Time to Response
Description: Time to response is defined as the number of days from the date of enrollment to the date of the first documented response of CR or PR. The median time to response will be summarized by descriptive statistics.
Time Frame: Up to 36 months
Population: No participants achieved an objective response, therefore a time to response could not be calculated.
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The disease control rate is defined as the best response recorded from the start of treatment including stable disease, until disease progression/recurrence (PD). Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, Complete Response (CR) is defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is defined as having at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is defined as having neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. The proportion of participants relative to the total size of the All Treated Subjects population having a demonstrated response of CR, PR, or SD, with a confirmatory scan will be reported.
Time Frame: Up to 36 months
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
proportion of participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0.21

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) is defined as the percentage of participants who achieved a best overall response of CR, PR and SD with a duration of response lasting at least 6 months or longer.
Time Frame: Up to 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
percentage of participants | 0

7. Secondary Outcome: Median Duration of Response
Description: The duration of response (DOR) will be calculated for participants who achieved a best overall response of CR or PR and calculated as the number of days from the date when CR or PR is first confirmed to the date of progression or death. Participants who do not have a documented progression or death will be censored on the last date of tumor assessment. The median DOR and 95% confidence intervals will be reported.
Time Frame: Up to 36 months
Population: No participants achieved an objective response, therefore a duration of response could not be calculated.
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 0

8. Secondary Outcome: Proportion of Participants With Reported Treatment-related Adverse Events (AEs)
Description: The proportion of participants with reported treatment-related adverse events, which are adverse events defined as having an attribution of possible, probable, or definite according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 4 will be reported.
Time Frame: Up to 36 months
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
Number analyzed (Participants) | 14
proportion of participants | 0.64

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Arm A: Tavo-EP, Pembrolizumab, Epacadostat
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tavo-EP, Pembrolizumab, Epacadostat (N=14)
Edema, Face (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) — Altered mental status
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood and lymphatic system disorders, Other (Blood and lymphatic system disorders) | 1 (1) — Aspiration of blood into airway due to disease progression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tavo-EP, Pembrolizumab, Epacadostat (N=14)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 2 (2)
Injection site reaction (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3) — Intermittent rash
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Nasuea (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Edema face (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Restless leg during evenings
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Tingling sensation in earlobe
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Discharge from tumor

LIMITATIONS AND CAVEATS:
The study closed earlier than expected during enrollment into Arm A. Arm B and Arm C were never opened to accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03823131/Prot_SAP_000.pdf